CLINICAL TRIAL: NCT04777981
Title: Efficacy of Cannabidiol in Combination With Red Algae (CBDRA60) to Prevent or Reduce Symptoms of COVID-19 and Post-Acute Sequelae of SARS-CoV-2 Infection PASC
Brief Title: (CBDRA60) to Prevent or Reduce Symptoms of COVID-19 and Prevention of Post-Acute Sequelae of SARS-CoV-2 Infection PASC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anewsha Therapeutics Inc. (Industry)
Collaborators: University of Michigan (Other); Biologics Consulting (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; SAR
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blind, placebo-controlled trial. Patients will be randomized to CBDRA60 supplement or placebo.
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBDRA60 supplement (Experimental): Daily sublingual tablet containing 30mg Cannabidiol and 30mg Red Algae, a total of 60mg per dose. Participants will take 2 tablets per day, sublingually and with food, taken approximately and at least, 8 hours apart, daily for 28 days. Participants will be mailed a supply of pills by an overnight courier service.
  Interventions: Dietary Supplement: CBDRA60 supplement
- Placebo (Placebo Comparator): Control subjects will receive daily oral placebo tablets of identical appearance and taste containing no CBDRA60.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CBDRA60 supplement — CBD is a non-psychotropic cannabinoid that has a broad spectrum of well-established anti-inflammatory and immunomodulatory effects. Red algae (Rhodophyta) are known for their potent anti-viral properties, non-toxicity and for being well tolerated in humans [15, 16]. Rhodophyta contain several sulfated polysaccharides that exhibit high antiviral activity against enveloped viruses.,
  Other Names: CBDRA60
  Arms: CBDRA60 supplement
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Coronavirus disease (COVID-19), caused by the novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), presents a major threat to human health. SARS-CoV-2 is highly infectious and is associated with extensive morbidity and mortality. Our study shares important features with other clinical trials using supplements or other widely available medications (e.g., Ascorbic Acid, Zinc, Vitamin D, Vitamin C). Our study shares two important elements with these previous studies, including:

1. The use of adaptive and cost-effective study design methods,
2. The testing of prophylactic supplementation using known, natural substances that have demonstrated safety and limited side effects.

The focus of this study is to use a supplement that combines Cannabidiol and Gigartina Red Algae in creating "CBDRA60", a sublingual tablet, which is hypothesized to help reduce the duration of symptoms in patients diagnosed with the novel coronavirus disease (COVID-19). The rationale and design of our trial (N=60), is as follows: 60 individuals newly diagnosed with COVID-19 infection will be randomized to one of two groups. They will either receive CBDRA60 (30mg CBD, 30mgRA / 60mg combo; 2x/daily with food or 120 mg total) or a placebo in a 1:1 ratio. The study duration will be 5 weeks. The primary outcome for newly diagnosed individuals is the prevention of disease progression which leads to hospitalization. The secondary outcome is a reduction in symptom severity scores.

COVID-19 patients with weakened innate immune systems may be susceptible to more severe disease and higher mortality. An impaired host immune response may lead to higher SARS-COV-2 viral load and subsequent overactivation of the adaptive immune system that results in cytokine release syndrome. CBD and Gigartina Red Algae can modulate both the innate and adaptive immune responses, have anti-viral activity and thereby can suppress the consequent hyperinflammatory response.

Viral infection activates a pathological inflammatory response to combat the pathogen and limit its spread. Viral pathogens, such as the severe acute respiratory syndrome (SARS) coronaviruses (SARS-CoV), and other viruses (such as HIV), have been linked to many human and animal diseases. Advancements in research over the past decade, has led to a better understanding of SARS-CoV biology and the mechanism by which this family of viruses, the coronaviridae, infect and enter the host cells (refs). SARS-CoV-2, a unique type of coronavirus, inhibits host defense by invading host cells, replicating, and infecting numerous tissues. Severe COVID-19 is associated with a cytokine storm, acute respiratory distress and consequent multiple organ pathology that can be fatal. This depictive storm is a result of increase in circulating levels of various proinflammatory cytokines including IL-6, IL-1 TNF-α as well as interferons (IFN-I; IFNα and IFNβ).

CBD CBD is a non-psychotropic cannabinoid that has a broad spectrum of well-established anti-inflammatory and immunomodulatory effects. For example, CBD administration in a murine model of lung injury, reduces lung inflammation through inhibition of immune cell cytokine production and suppression of leukocyte infiltration. Our premise is that similar CBD-induced effects would be highly applicable and hugely beneficial to mitigating the acute respiratory distress syndrome observed in COVID-19. Published evidence also indicates that CBD can inhibit viral replication. Red algae (Rhodophyta) are known for their potent anti-viral properties, non-toxicity and for being well tolerated in humans. Rhodophyta contain several sulfated polysaccharides that exhibit high antiviral activity against enveloped viruses, including important human pathogens such as herpes simplex virus (HSV), human cytomegalovirus, dengue virus and respiratory syncytial virus. Sulfated polysaccharides can exert their anti-viral effects through interacting with the external glycoprotein of the virion envelope preventing attachment of the virus to cell surface receptors. Red algae also contain mannose specific lectins that specifically interact with viral envelope glycoproteins including the spike glycoprotein specific to SARS-CoV2 to inhibit viral entry.

It is our premise that by using a safe and tolerable dose of the formulated CBDRA60 sublingual tablet, participants could either be protected from viral infection of the SARS-CoV-2 virus (COVID-19) or in subjects that are already infected, CBDRA60, could prevent virus attachment, mitigate virus-induced inflammation and avoid a cytokine storm, enabling a faster recovery.

DETAILED DESCRIPTION:
The trial is a randomized, double blind, placebo-controlled trial with a total of 60 participants located in the state of Michigan. Patients will be randomized to CBDRA60 supplement or placebo.

All participants will be newly diagnosed as positive for SARS-CoV2 (assessed using a PCR test).

Each participant will be randomized to either CBDRA60 or placebo in a 1:1 ratio. The study duration for each participant will be 5 weeks, including taking the supplementation (active or placebo for 28 days). Of the 60 participants, 30 participants will receive CBDRA60 and 30 participants will receive the placebo. The infected individuals will be followed to assess disease progression defined as the need for hospitalization.

For participants receiving the CBDRA60 supplementation, it aims to reduce

1. The need to be hospitalized and
2. Self-reported disease severity and resolution over 5 weeks Participants will self-report symptom severity and disease progression through weekly questionnaires. For each specified COVID-19 related symptom (fever, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea), participants will report one of the following 3 options: none (score of 0), mild (score of 1), moderate (score of 2) or severe (score of 3) except for new loss of taste or smell which will be assessed using a binary score (0 = no loss of taste/smell, 1 = loss of taste/smell) in accordance with the HHS guidelines (Sep 2020 document). The total disease severity score will be the average across all potential symptoms. The escalation protocol for any participants that experience symptoms that are more than mild or continue to progress will be directed to contact their primary care physician or their appropriate emergency care facility.

Supplementation Daily sublingual tablet containing 30mg Cannabidiol and 30mg Red Algae, a total of 60mg per dose. Participants will take 2 tablets per day, sublingually and with food, taken approximately and at least, 8 hours apart, daily for 28 days. Participants will be mailed a supply of pills by an overnight courier service.

Control subjects will receive daily oral placebo tablets of identical appearance and taste containing no CBDRA60.

Study procedures Recruitment Participants will be recruited across Michigan via social media; community advocacy groups and equity initiatives; flyers and electronic communications distributed in healthcare centers, COVID-19 testing centers, and other avenues. Recruitment will primarily be conducted remotely and prospective participants will be asked to complete a web-based HIPAA-secure screening survey by the MB Clinical or VSafe system. Screen-eligible participants will be contacted by phone by research staff to complete the screening process using on-line consent forms.

Baseline and follow-up Participants will receive messages as a reminder to take study pills. They will also be instructed to complete 1x per week online questionnaires for 5 weeks and an additional post study follow-up questionnaire at week 8. The questionnaire will include items on adherence with randomized supplementation with CBDRA60/placebo, use of non-trial supplements of CBD, development of symptoms and new illness, and self-report of disease progression and severity status. Non-responders to online notification will be telephoned to collect study data.

Data Management Using ClinOne or VSafe Platform

ClinOne, a clinical research organization (CRO) with a Vsafe platform will be implemented for key areas of improvement of patient engagement and retention throughout the investigation. It provides remote online services between patients and the clinicians in charge. It further provides services for:

* Required screening criteria,
* Questionnaires,
* Study contact,
* Recorded investigatory meetings,
* CEO and KOL presentation and important messages,
* Training videos. All through a secure online platform.

All the services can be accessed via the ClinOne or VSafe platform. Patients will use the platform for reminders, to access study information, report questions or concerns, and communicate with principal investigators and physician. The platform allows the clinical trial leader to schedule events via its manager system (S.O.E.M). It is a secure portal to share approved study documents, provide a concierge and knowledge digital base, research visits, and ePro lite which will be used to deliver the questionnaires to patients and guarantee the collection of evaluable data. For reminders on when to take the CBDRA 60 sublingual tablet an electronic eDosing adherence reminder will be available to notify the study participants.

Lastly, in order to monitor the subjects health, remotely, and to collect additional biometric data, a smart BioIntelliSense's BioButton™ medical-grade device and HIPAA-compliance data service will be used. This enables effortless remote, multi-parameter data capturing that measures vital signs in real time. It comprises a single disposable on-body sensor for continuous monitoring of temperature, oximeter readings, respiratory rate, heart rate at rest, body position, sleep and activity state for 90-days. Alternatively, a similar oximeter / thermometer combination will be provided.

Assessed symptoms are Fever, Cough, Shortness of Breath, Fatigue, Muscle or body aches, Headache, New loss of taste, New loss of smell, Congestion or runny nose, Nausea, Vomiting, Diarrhea. Each patient will have a composite score ranging from 0-36/day.

1. Symptom Resolution: Fever [Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of fever based on a 0-3 scale: 0 = ≤98.6oF, 1 = >98.6 oF - 100.4 oF, 2 = > 100.4 oF - 102.6 oF, 3 = >102.6 oF
2. Symptom Resolution: Cough [Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of cough based on a 0-2 scale: 0 = no cough, 1 = mild/moderate, 2 = severe (How does the individual discriminate between mild and moderate?)
3. Symptom Resolution: Shortness of Breath [Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of shortness of breath based on a 0-3 scale: 0 = no shortness of breath, 1 = with moderate intensity exercise 2 = with walking on flat surface 3 = short of breath with getting dressed or daily activities
4. Symptom Resolution: Fatigue [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of fatigue based on a 0-3 scale:) 0=no fatigue, 1=mild fatigue, 2=moderate fatigue, 3=severe fatigue.
5. Symptom Resolution: Muscle/body aches [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of muscle/body aches based on a 0-3 scale: 0=no muscle/body aches, 1=mild muscle/body aches, 2=moderate muscle/body aches , 3=severe muscle/body aches.
6. Symptom Resolution: Headache [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of headache based on a 0-3 scale: 0=no headache, 1=mild headache, 2=moderate headache, 3=severe headache.
7. Symptom Resolution: New loss of taste [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of new loss of taste based on a binary scale: 0=no loss of taste, 1= loss of taste.

   Symptom Resolution: New loss of smell [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of new loss of smell based on a binary scale: 0=no loss of smell, 1= loss of smell.
8. Symptom Resolution: Congestion/ runny nose [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of congestion/runny nose on a 0-3 scale: 0=no congestion/runny nose, 1=mild congestion/runny nose , 2=moderate congestion/runny nose , 3=severe congestion/runny nose .
9. Symptom Resolution: Nausea [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of nausea on a 0-3 scale:0=no nausea, 1=mild nausea, 2=moderate nausea, 3=severe nausea.
10. Symptom Resolution: Vomiting [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of vomiting on a 0-3 scale: 0=no vomiting, 1=mild vomiting, 2=moderate vomiting, 3=severe vomiting.
11. Symptom Resolution: Diarrhea [ Time Frame: 35 days] The number of days required to reach a score of 0 from the symptom category of diarrhea on a 0-3 scale: 0=no diarrhea, 1=mild diarrhea, 2=moderate diarrhea, 3=severe diarrhea.
12. Day 28 Composite Symptoms [ Time Frame: 35 days] Total symptom composite score at day 5 of study supplementation: Symptom categories of fever based on a 0-3 scale: 0 = ≤98.6 oF, 1 = >98.6- 100.6 oF, 2 = > 100.6 - 102.6 oF, 3 = >102 oF; Cough on a 0-3 scale: 0 = no cough, 1 = mild, 2 = moderate, 3 = severe; Shortness of Breath on a 0-3: 0 = no shortness of breath, 1 = with moderate intensity exercise 2 = with walking on flat surface 3 = short of breath with getting dressed or daily activities; and Fatigue on a 0-3 scale: 0 = No fatigue/energetic, 1=mild fatigue, 2=moderate fatigue, 3=severe fatigue.
13. Hospitalizations/ER visits [ Time Frame: 35 days] Differences in hospitalization, ER visits, mortality events between the study arms
14. Severity of Symptoms [Time Frame: 35 days] Differences in severity of symptoms between study arms
15. Adjunctive Medications [ Time Frame: 35 days] Differences in number of patients who were prescribed adjunctive medications for their diagnosis between study arms
16. Supplementation Side Effects [ Time Frame: 35 days] Differences in number of patients in study arms who experienced side effects from the supplements.

ELIGIBILITY:
Inclusion Criteria:

The study population will include individuals who tested positive for COVID-19 infection based on a PCR test. The study population is defined as adults ≥ 18 years of age with no comorbidities and absence of pre-existing conditions (see exclusion criteria below).

* Baseline drug screen for schedule 1 narcotics
* All participants are required to understand and provide informed consent before any assessment is performed
* Be willing and able to complete an online questionnaire
* Be able to understand and agrees to comply with planned study procedures and be available for all study visits
* Participants who have received the Pfizer or Moderna vaccine are allowed to be enrolled in study if they have a PCR positive test

Exclusion Criteria:

* Current hospitalization
* Participation in any other COVID-19 trial
* Individuals that are taking antiviral medications
* Baseline lab/drug screen shows consumption of a schedule 1 narcotic
* Prior diagnosis of cancer and currently undergoing radiation, chemotherapy, or immunotherapy; excluding basal cell skin carcinoma
* Participants who have been diagnosed as HIV positive or taking anti-HIV therapy
* Female participants who are pregnant or breastfeeding, lactating, or planning a pregnancy during the trial.
* Female subjects who is/are breastfeeding or plans to breastfeed
* Medical disease or conditions such as high-risk comorbidities such as: diabetes, chronic obstructive pulmonary disease (COPD) or emphysema, history of heart attack or stroke, history of coronary bypass surgery or coronary angioplasty or stent, history of hospitalization for heart failure, etc.
* Demonstrated inability to comply, tell the truth (as defined by PI, study investigator on subjects health condition) with the study procedures
* History of hypersensitive or severe allergic reactions
* Anticipated need for immunosuppressive treatment within the next 6 months
* Received immunoglobulins and or any blood or blood products within the 4 months of being enrolled in this investigation
* Blood dyscrasias or significant disorder of coagulation.
* Severe Liver disease including chronic liver disease, fatty liver, cirrhosis or awaiting transplant.
* History of alcohol abuse or other recreational drug abuse of schedule 1 narcotics within 6 months of being enrolled in the study.
* Subjects diagnosed with:

  * Kidney disease (CKD) | End-Stage Renal Disease (ESRD) or dialysis.
  * A history of Calcium Oxalate kidney stones
  * Mineral bone disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-05 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Decreased hospitalization | 35 days
  Number of participants hospitalized and/or requiring repeat emergency room visit from COVID-19 related complications.

SECONDARY OUTCOMES:
Resolution of COVID-19 symptoms | 35 days
  Time at which the patient is completely symptom free. Number of days to reach a 30-50 percent change in the cumulative 0-36 symptom score with each symptom evaluated on a 0-3 scale. Lower is better, higher is worse Assessed symptoms are Fever, Cough, Shortness of Breath, Fatigue, Muscle or body aches, Headache, New loss of taste, New loss of smell, Congestion or runny nose, Nausea, Vomiting, Diarrhea. Each patient will have a composite score ranging from 0-36/day.
  Example symptom resolution: Shortness of Breath [Time Frame: 35 days] Number of days required to reach a score of 0 from the symptom category of shortness of breath based on a 0-3 scale: 0 = no shortness of breath, 1 = with moderate intensity exercise 2 = with walking on flat surface 3 = short of breath with getting dressed or daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Stylianou, PHD, Principal Investigator — Anewsha Therapeutics
Locations (1):
- Anewsha Therapeutics / Comco R&D, Hanover, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fauci AS, Lane HC, Redfield RR. Covid-19 - Navigating the Uncharted. N Engl J Med. 2020 Mar 26;382(13):1268-1269. doi: 10.1056/NEJMe2002387. Epub 2020 Feb 28. No abstract available. PMID 32109011
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Wang R, DeGruttola V, Lei Q, Mayer KH, Redline S, Hazra A, Mora S, Willett WC, Ganmaa D, Manson JE. The vitamin D for COVID-19 (VIVID) trial: A pragmatic cluster-randomized design. Contemp Clin Trials. 2021 Jan;100:106176. doi: 10.1016/j.cct.2020.106176. Epub 2020 Oct 10. PMID 33045402
- [Background] Miranda-Massari JR, González MJ, Marcial-Vega VA, Soler JD: A Possible Role for Ascorbic Acid in COVID-19. Journal of Restorative Medicine 2020, 10.
- [Background] Bauer SR, Kapoor A, Rath M, Thomas SA. What is the role of supplementation with ascorbic acid, zinc, vitamin D, or N-acetylcysteine for prevention or treatment of COVID-19? Cleve Clin J Med. 2020 Jun 8. doi: 10.3949/ccjm.87a.ccc046. Online ahead of print. PMID 32513807
- [Background] Skalny AV, Rink L, Ajsuvakova OP, Aschner M, Gritsenko VA, Alekseenko SI, Svistunov AA, Petrakis D, Spandidos DA, Aaseth J, Tsatsakis A, Tinkov AA. Zinc and respiratory tract infections: Perspectives for COVID-19 (Review). Int J Mol Med. 2020 Jul;46(1):17-26. doi: 10.3892/ijmm.2020.4575. Epub 2020 Apr 14. PMID 32319538
- [Background] Shi Y, Wang Y, Shao C, Huang J, Gan J, Huang X, Bucci E, Piacentini M, Ippolito G, Melino G. COVID-19 infection: the perspectives on immune responses. Cell Death Differ. 2020 May;27(5):1451-1454. doi: 10.1038/s41418-020-0530-3. Epub 2020 Mar 23. No abstract available. PMID 32205856
- [Background] Huestis MA. Human cannabinoid pharmacokinetics. Chem Biodivers. 2007 Aug;4(8):1770-804. doi: 10.1002/cbdv.200790152. No abstract available. PMID 17712819
- [Background] Vaninov N. In the eye of the COVID-19 cytokine storm. Nat Rev Immunol. 2020 May;20(5):277. doi: 10.1038/s41577-020-0305-6. No abstract available. PMID 32249847
- [Background] Ragab D, Salah Eldin H, Taeimah M, Khattab R, Salem R. The COVID-19 Cytokine Storm; What We Know So Far. Front Immunol. 2020 Jun 16;11:1446. doi: 10.3389/fimmu.2020.01446. eCollection 2020. PMID 32612617
- [Background] Lee JS, Shin EC. The type I interferon response in COVID-19: implications for treatment. Nat Rev Immunol. 2020 Oct;20(10):585-586. doi: 10.1038/s41577-020-00429-3. PMID 32788708
- [Background] Pellati F, Borgonetti V, Brighenti V, Biagi M, Benvenuti S, Corsi L. Cannabis sativa L. and Nonpsychoactive Cannabinoids: Their Chemistry and Role against Oxidative Stress, Inflammation, and Cancer. Biomed Res Int. 2018 Dec 4;2018:1691428. doi: 10.1155/2018/1691428. eCollection 2018. PMID 30627539
- [Background] Ribeiro A, Almeida VI, Costola-de-Souza C, Ferraz-de-Paula V, Pinheiro ML, Vitoretti LB, Gimenes-Junior JA, Akamine AT, Crippa JA, Tavares-de-Lima W, Palermo-Neto J. Cannabidiol improves lung function and inflammation in mice submitted to LPS-induced acute lung injury. Immunopharmacol Immunotoxicol. 2015 Feb;37(1):35-41. doi: 10.3109/08923973.2014.976794. Epub 2014 Oct 30. PMID 25356537
- [Background] Wang J, Hajizadeh N, Moore EE, McIntyre RC, Moore PK, Veress LA, Yaffe MB, Moore HB, Barrett CD. Tissue plasminogen activator (tPA) treatment for COVID-19 associated acute respiratory distress syndrome (ARDS): A case series. J Thromb Haemost. 2020 Jul;18(7):1752-1755. doi: 10.1111/jth.14828. Epub 2020 May 11. PMID 32267998
- [Background] Nakashima H, Kido Y, Kobayashi N, Motoki Y, Neushul M, Yamamoto N. Antiretroviral activity in a marine red alga: reverse transcriptase inhibition by an aqueous extract of Schizymenia pacifica. J Cancer Res Clin Oncol. 1987;113(5):413-6. doi: 10.1007/BF00390034. PMID 2442171
- [Background] Bourgougnon N, Lahaye M, Quemener B, Chermann J, Rimbert M, Cormaci M, Furnari G, Kornprobst J: Annual variation in composition andin vitro anti-HIV-1 activity of the sulfated glucuronogalactan fromSchizymenia dubyi (Rhodophyta, Gigartinales). Journal of applied phycology 1996, 8:155-161
- [Background] Bouhlal R, Haslin C, Chermann JC, Colliec-Jouault S, Sinquin C, Simon G, Cerantola S, Riadi H, Bourgougnon N. Antiviral activities of sulfated polysaccharides isolated from Sphaerococcus coronopifolius (Rhodophytha, Gigartinales) and Boergeseniella thuyoides (Rhodophyta, Ceramiales). Mar Drugs. 2011;9(7):1187-1209. doi: 10.3390/md9071187. Epub 2011 Jul 6. PMID 21822410
- [Background] Duarte ME, Noseda DG, Noseda MD, Tulio S, Pujol CA, Damonte EB. Inhibitory effect of sulfated galactans from the marine alga Bostrychia montagnei on herpes simplex virus replication in vitro. Phytomedicine. 2001 Jan;8(1):53-8. doi: 10.1078/0944-7113-00007. PMID 11292240
- [Background] Zhu W, Chiu LC, Ooi VE, Chan PK, Ang PO Jr. Antiviral property and mode of action of a sulphated polysaccharide from Sargassum patens against herpes simplex virus type 2. Int J Antimicrob Agents. 2004 Sep;24(3):279-83. doi: 10.1016/j.ijantimicag.2004.02.022. PMID 15325432
- [Background] Mazumder S, Ghosal PK, Pujol CA, Carlucci MJ, Damonte EB, Ray B. Isolation, chemical investigation and antiviral activity of polysaccharides from Gracilaria corticata (Gracilariaceae, Rhodophyta). Int J Biol Macromol. 2002 Dec 20;31(1-3):87-95. doi: 10.1016/s0141-8130(02)00070-3. PMID 12559431
- [Background] Pujol CA, Carlucci MJ, Matulewicz MC, Damonte EB: Natural sulfated polysaccharides for the prevention and control of viral infections. In Bioactive Heterocycles V. Springer; 2007: 259-281
- [Background] Sato Y, Morimoto K, Kubo T, Sakaguchi T, Nishizono A, Hirayama M, Hori K. Entry Inhibition of Influenza Viruses with High Mannose Binding Lectin ESA-2 from the Red Alga Eucheuma serra through the Recognition of Viral Hemagglutinin. Mar Drugs. 2015 May 29;13(6):3454-65. doi: 10.3390/md13063454. PMID 26035023
- [Background] Singh RS, Walia AK. Lectins from red algae and their biomedical potential. J Appl Phycol. 2018;30(3):1833-1858. doi: 10.1007/s10811-017-1338-5. Epub 2017 Nov 20. PMID 32214665
- [Background] Hirayama M, Shibata H, Imamura K, Sakaguchi T, Hori K. High-Mannose Specific Lectin and Its Recombinants from a Carrageenophyta Kappaphycus alvarezii Represent a Potent Anti-HIV Activity Through High-Affinity Binding to the Viral Envelope Glycoprotein gp120. Mar Biotechnol (NY). 2016 Feb;18(1):144-60. doi: 10.1007/s10126-015-9677-1. Epub 2015 Nov 23. PMID 26593063
- [Background] Barre A, Damme EJMV, Simplicien M, Benoist H, Rouge P. Man-Specific, GalNAc/T/Tn-Specific and Neu5Ac-Specific Seaweed Lectins as Glycan Probes for the SARS-CoV-2 (COVID-19) Coronavirus. Mar Drugs. 2020 Oct 29;18(11):543. doi: 10.3390/md18110543. PMID 33138151